CLINICAL TRIAL: NCT00733278
Title: Acceptability and Technical Feasibility of Insertion of a Copper IUD at Time of Elective C-section: A Pilot Study
Brief Title: Intrauterine Contraceptive Device (IUD) Placement at Time of C-Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12670-01
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-07

CONDITIONS: Contraception
Keywords: Postpartum contraception; Copper IUD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Copper IUD (Experimental): Copper IUD
  Interventions: Device: Copper IUD ( ParaGard Intrauterine Contraceptive Device)

INTERVENTIONS:
Device: Copper IUD ( ParaGard Intrauterine Contraceptive Device) — Intraoperative placement of copper IUD at time of C-section
  Other Names: ParaGard Intrauterine Contraceptive Device

SUMMARY:
This is a pilot study of up to 10 women, which will test the hypothesis that the placement of copper IUDs through the uterine incision at the time of uncomplicated elective C-section is technically feasible and acceptable to women seeking long-term contraception.

DETAILED DESCRIPTION:
Women will be enrolled in this study during late prenatal care. Consent for placement of the IUD will be verified prior to elective C-section. After removal of the placenta, the copper IUD will be placed through the incision at the fundus and the tail strings will be delivered through the cervix. Data will be collected about patient bleeding and possible infection during the immediate postoperative period. The visibility of the strings will be verified at discharge and at 2 and 6 weeks postpartum. Fundal placement of the IUD will be verified by ultrasound at the patient's last visit.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Requires elective C-section
* Desires long-term contraception

Exclusion Criteria:

* Contraindications to copper IUD

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita L Nelson, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles BRI, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women in prenatal clinic were approached in the third trimester if they were to be scheduled for elective C-section. If they were interested in using Copper IUD, their informed consent was obtained. At the time of elective C-section, their continued interest in study participation was verified.
Groups:
- Copper IUD: Women undergoing elective C-section who request long-term contraception with Copper IUD.
Period: Overall Study
Arm/Group | Copper IUD
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IUD Placement
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Data not relevant to analysis, and, therefore, not collected.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Successful Retention of IUD
Time Frame: 6 weeks
Measure: Number; unit: participants
Groups:
- IUD Placement: IUD placement following removal of placenta at time of elective C-section
Arm/Group | IUD Placement
Number analyzed (Participants) | 7
participants | 7

2. Secondary Outcome: Visibility Within the Vagina of IUD Strings at All Times.
Time Frame: At 3 days, 2 weeks and 6 weeks postpartum
Measure: Number; unit: participants
Groups:
- IUD Strings: Visibility of IUD strings within the vagina at all times.
Arm/Group | IUD Strings
Number analyzed (Participants) | 7
participants | 7

ADVERSE EVENTS:
Arm/Group | Copper IUD
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Pilot study involving only seven subjects, which limits generalizability of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No